CLINICAL TRIAL: NCT07355335
Title: A Phase 1 Study of Menin-KMT2A Inhibitor Ziftomenib (KO-539) in Combination With Cereblon E3 Ligase Modulator Mezigdomide (CC-92480) in Adolescents and Adults With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Ziftomenib + Mezigdomide in Adolesc. and Adults w/ R/R AML
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Kura Oncology, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Amir Fathi, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-804
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: KMT2A-rearranged; NPM1-mutant Refractory or Relapsed AML
Keywords: KMT2A rearrangement; NPM1c mutation; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ziftomenib and Mezigdomide (Experimental): Ziftomenib will be taken orally once daily of each cycle. A drug diary will be provided to participants to document information about taking ziftomenib.
  Mezigdomide will be taken orally once daily on days 1-21 or possibly days 1-14 of each cycle. The study doctor will confirm which days mezigdomide will be taken on. A drug diary will be provided to participants to document information about taking mezigdomide.
  Interventions: Drug: Ziftomenib; Drug: Mezigdomide

INTERVENTIONS:
Drug: Ziftomenib — Capsule taken orally once daily on days 1-28 of each 28-day cycle.
  Other Names: KO-539
Drug: Mezigdomide — Capsule taken orally once daily on days 1-21 or possibly days 1-14 of each 28-day cycle.
  Other Names: BMS-986348; CC-92480

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of mezigdomide in combination with ziftomenib in adolescent and adult participants with either KMT2A-rearranged (KMT2A-r) or NPM1-mutant relapsed or refractory acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved ziftomenib and mezigdomide as a treatment for any disease.

Duration of treatment will depend on individual response, evidence of disease progression, and tolerance. The total treatment period will be 12 cycles. If you have completed treatment, you will be followed of up to 12 months. If you do not, complete treatment, you will be followed for 30 days after discontinuation of treatment.

It is expected that about 24 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years during dose escalation portion of study, patients must weigh ≥40 kg.
* Age >12 years during dose expansion portion of study, patients must weight ≥40 kg.
* Diagnosis of AML per the WHO Classification of Hematolymphoid Tumors (5th Edition) with documented KMT2A rearrangement or NPM1 cytoplasmic-type (NPM1c) mutation. KMT2A-rearrangements must be confirmed by FISH or RNA-based fusion calling by a CLIA-certified laboratory. This study will only enroll KMT2A gene rearrangements in which there is a translocation between the N-terminal portion of KMT2A and a fusion partner, and will not include KMT2A partial tandem duplications (PTDs) or other structural alterations of KMT2A. NPM1c mutations must be confirmed by DNA sequencing in a CLIA-certified laboratory. Patients with myeloid sarcoma are eligible only if concurrent bone marrow involvement is present. Patients must have at least 5% bone marrow disease by morphology at the time of study entry.
* Patients with NPM1 mutated AML must either be FLT3 ITD wild type or have an ITD allelic ratio of <0.05 (i.e. not eligible for a targeted FLT3 tyrosine kinase inhibitor).
* Patients must have relapsed or be refractory to at least one prior line of conventional therapy for AML or MDS-AML.
* Eastern Cooperative Oncology Group (ECOG) performance status must be 0, 1, or 2; Karnofsky ≥50 for patients ≥16 years of age; and Lansky ≥50 for patients ≥12 to 16 years of age.
* Participants must meet the following organ and marrow function as defined below:

  * Leukocytes <25,000/mcL (hydroxyurea, leukapheresis, or single dose of cytarabine 1 g IV are permitted to meet this criterion)
  * AST(SGOT)/ALT(SGPT) ≤5 × institutional ULN and total bilirubin ≤ 2x institutional ULN unless related to leukemic involvement or known Gilbert's syndrome (for bilirubin).
  * Cardiac LVEF of ≥40%, as measured by echocardiogram or MUGA scan
  * Glomerular filtration rate (GFR)≥30 mL/min/1.73 m2
* The patient, a parent (if the patient is <18 years old), or a legally authorized representative must be able to understand and provide informed consent.
* Patients of childbearing potential are eligible for the study but must comply with the pregnancy prevention plan for study drugs. See Appendix B for details.
* Patient's life expectancy attributed to AML must be greater than 3 months.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Life expectancy attributed to malignancy other than AML must be greater than 24 months. Patients with concurrent malignancy who are receiving chemotherapy or whose disease is uncontrolled or progressing are not eligible.

Exclusion Criteria:

* AML diagnosis without KMT2A-rearrangement or NPM1-mutation. KMT2A-PTD patients and patients with KMT2A alterations other than translocations are excluded.
* Active central nervous system (CNS) involvement by AML (i.e., CNS-2 or CNS-3 disease). Previously treated CNS disease or those receiving prophylactic intrathecal chemotherapy per institutional standard is allowed.
* Myeloid sarcoma or extramedullary disease without bone marrow disease.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1 by the NCI-CTCAE version 5.0) with the exception of alopecia.
* Participants who are receiving any other investigational agents for this condition.
* Clinically active HIV disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to mezigdomide (i.e. lenalidomide, thalidomide)
* Patient received chemotherapy, immunotherapy, radiation therapy, or ancillary therapy that is considered to be investigational <7 days prior to the first dose of ziftomenib and mezigdomide, or within 5 drug half-lives prior to the first dose of study drug, whichever is longer.
* Patients with psychiatric, familial, or geographic factors that may impede ability to provide informed consent, to follow study protocol, or hamper study compliance.
* Any other significant medical or psychosocial comorbidities that would preclude the patient from participating in the study or would confound interpretation of study results.
* Patients with the following uncontrolled comorbidities will be excluded: symptomatic congestive heart failure (NYHA class 3 or higher), unstable angina pectoris, serious cardiac arrhythmia as uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia (type 1 NSTEMI), active, uncorrected conduction abnormalities as Mobitz 2 or third degree heart block (not excluded if pacemaker placed), myocardial infarction with evidence of residual abnormalities within 6 months prior to enrollment. An elevation in troponin is not an exclusion criterion if there are no evidence of residual cardiac dysfunction or ongoing ischemic event. Patients with congenital conduction abnormalities as Wolff-Parkinson White, long QT syndrome, or Brugada syndrome may be eligible with consultation of cardiology confirming stability.
* Mean corrected QT interval corrected for heart rate by Frederica's formula (QTcF)>480ms.
* Patients on dialysis.
* Patients with active infection that are deemed controlled will be permitted to enroll. Patients with uncontrolled infection may enroll once infection is treated and brought under control.
* Subjects who have undergone a hematopoietic stem cell transplant (HSCT) within 90 days of the first dose of treatment on study, or subjects on immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD), requiring an equivalent dose of ≥ 0.5mg/kg/day of prednisone or therapy beyond systemic corticosteroids. (The use of topical steroids for ongoing skin GVHD is permitted.)
* Patients who are unable to swallow pills.
* Patient with gastrointestinal disease or surgery (e.g., gastric bypass surgery) that may significantly alter the absorption of mezigdomide and/or other oral study treatment.
* Proton pump inhibitors and potassium-competitive acid blockers are not permitted due to limited absorption of mezigdomide if the stomach is not acidic; a 7-day washout is required prior to start of study treatment.
* Has active Hepatitis B or C

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-07-09 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the start of treatment until participant withdrawal, death, or removal from study, whichever comes first, assessed up to 2 years after initial dose of study treatment.
  To characterize the safety and tolerability of mezigdomide in combination with ziftomenib, all reported toxicities will be summarized by toxicity type and maximum grade and will be reported as numbers and percentages. All participants who receive at least one dose of study treatments will be evaluable for toxicity.
Recommended phase 2 dose (RP2D) of mezigdomide in combination with ziftomenib. | From start of treatment to end of 12 cycles (each cycle is 28 days).
  The RP2D of mezigdomide in combination with ziftomenib will be determined in the dose escalation phase via a traditional 3+3 dose escalation design.

SECONDARY OUTCOMES:
Complete remission/complete remission with partial hematologic recovery (CR/CRh) and overall response rate (ORR) | From start of treatment to end of 12 cycles (each cycle is 28 days) or until participant withdrawal, death, or removal from study, whichever comes first.
  CR/CRh rate and overall response rate will be summarized using point estimates and exact binomial 90% confidence intervals in patients treated with RP2D.
2-year overall and relapse-free survival rates | From the start of treatment until participant withdrawal, death, or removal from study, whichever comes first, assessed up to 2 years after initial dose of study treatment.
  Two-year overall survival and relapse-free survival will be estimated using the Kaplan-Meier method with 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Fathi, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Amir Fathi, MD (AFATHI@mgh.harvard.edu) at 617-724-1124. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation